CLINICAL TRIAL: NCT01428830
Title: Non-inferiority of Short-term Catheterization Following Fistula Repair Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EngenderHealth (Other)
Collaborators: World Health Organization (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A65783
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Vaginal Fistula
Keywords: fistula; catheter; surgery; obstetrics; gynecology; urology
MeSH Terms: conditions — Vaginal Fistula; Fistula | interventions — Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 7-day catheterization (Experimental)
  Interventions: Procedure: 7-day catheterization following fistula repair surgery
- 14-day catheterization (Active Comparator)
  Interventions: Procedure: 14 day catheterization

INTERVENTIONS:
Procedure: 7-day catheterization following fistula repair surgery — This group will have an indwelling urethral catheter for 7 days following fistula repair surgery.
  Arms: 7-day catheterization
Procedure: 14 day catheterization — This group will have an indwelling urethral catheter for 14 days following fistula repair surgery.
  Arms: 14-day catheterization

SUMMARY:
This facility-based, multi-center randomized controlled trial (RCT) will test the non-inferiority of short-term (7 day) urethral catheterization compared to longer-term (14 day) urethral catheterization in terms of predicting fistula repair breakdown three months following urinary fistula repair surgery. The study will be conducted among 507 women with simple fistula presenting at 8 study sites in Sub-Saharan Africa for fistula repair surgery.

DETAILED DESCRIPTION:
A vaginal fistula is a devastating condition, affecting an estimated 2 million girls and women across Africa and Asia. Finding ways of providing services in a more efficient and cost-effective manner, without compromising surgical outcomes and the overall health of the patient, is paramount. Shortening the duration of urethral catheterization following fistula repair surgery would increase treatment capacity (by freeing available bed space and increasing availability of nursing staff), lower costs of services, and potentially lower risk of healthcare-associated infections among fistula patients. There is a lack of empirical evidence supporting any particular length of time for urethral catheterization following fistula repair surgery.

This facility-based, multi-center randomized controlled trial (RCT) will test the non-inferiority of short-term (7 day) urethral catheterization compared to longer-term (14 day) urethral catheterization in terms of predicting fistula repair breakdown. The primary outcome is fistula repair breakdown three months following fistula repair surgery as assessed by a urinary dye test, a routine practice in fistula repair services. t. Secondary outcomes will include repair breakdown one week following catheter removal, intermittent catheterization due to urinary retention and the occurrence of septic or febrile episodes, prolonged hospitalization (defined as a stay at the facility beyond one week following initial catheter removal related to an adverse event), catheter blockage, and self-reported residual incontinence. This study will be conducted among 507 women with simple fistula presenting at 8 study sites for fistula repair surgery over the course of 16-18 months at each site.

ELIGIBILITY:
Inclusion Criteria:

* Have a "simple" fistula, as determined at the end of fistula repair surgery (irrespective of the number of prior repair attempts and the cause of the fistula, with the exceptions noted under the exclusion criteria below)
* Have a closed fistula at completion of surgery
* Have a closed fistula 7 days after surgery (i.e. at the time of randomization)
* Understand study procedures and requirements
* Agree to return to the facility for one follow-up visit three month after the date of surgery
* Provide informed consent to participate in the study or in the case of non-emancipated minors, both consent to the study and receive proxy consent to participate in the study
* Have no contraindications precluding their participation.

Exclusion Criteria:

* Have a fistula that is determined to be "not simple" (i.e. intermediate or complex)
* Have a fistula that is radiation-induced, associated with cancer or due to lymphogranuloma venereum (These cases will be excluded because the healing process is very different from fistula resulting from other causes. We expect there to be few cases of these fistulas at the study sites)
* Have a fistula that is not closed immediately after surgery or 7 days after surgery (i.e. at the time of randomization)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Fistula repair breakdown three months following fistula repair surgery as assessed by a urinary dye test. | 3 months

SECONDARY OUTCOMES:
Repair breakdown one week following catheter removal | 14 days or 21 days post-repair
Intermittent catheterization due to urinary retention | 7 or 14 days post repair
Prolonged hospitalization | 14 or 21 days post-repair
Catheter blockage | 14 or 21 days post repair
Self-reported residual incontinence | 3 months
The occurrence of septic or febrile episodes | 14 or 21 days post-repair

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Barone, DVM, MS, Principal Investigator — EngenderHealth; Mariana Widmer, Study Director — World Health Organization
Locations (8):
- Hôpital Saint Joseph, Kinshasa, Democratic Republic of the Congo
- Gondar University Hospital, Gonder, Ethiopia
- L'Hôpital Préfectoral de Kissidougou, Kissidougou, Guinea
- Kenyatta National Hospital, Nairobi, Kenya
- National Obstetric Fistula Centre, Abakaliki, Nigeria
- Maternité Centrale de Zinder, Zinder, Niger
- Aberdeen Women's Centre, Freetown, Sierra Leone
- Kagando Hospital, Kasese District, Uganda

REFERENCES:
- [Derived] Barone MA, Widmer M, Arrowsmith S, Ruminjo J, Seuc A, Landry E, Barry TH, Danladi D, Djangnikpo L, Gbawuru-Mansaray T, Harou I, Lewis A, Muleta M, Nembunzu D, Olupot R, Sunday-Adeoye I, Wakasiaka WK, Landoulsi S, Delamou A, Were L, Frajzyngier V, Beattie K, Gulmezoglu AM. Breakdown of simple female genital fistula repair after 7 day versus 14 day postoperative bladder catheterisation: a randomised, controlled, open-label, non-inferiority trial. Lancet. 2015 Jul 4;386(9988):56-62. doi: 10.1016/S0140-6736(14)62337-0. Epub 2015 Apr 21. PMID 25911172
- [Derived] Barone MA, Frajzyngier V, Arrowsmith S, Ruminjo J, Seuc A, Landry E, Beattie K, Barry TH, Lewis A, Muleta M, Nembunzu D, Olupot R, Sunday-Adeoye I, Wakasiaka WK, Widmer M, Gulmezoglu AM. Non-inferiority of short-term urethral catheterization following fistula repair surgery: study protocol for a randomized controlled trial. BMC Womens Health. 2012 Mar 20;12:5. doi: 10.1186/1472-6874-12-5. PMID 22433581